CLINICAL TRIAL: NCT05486091
Title: A Feasibility Open Trial of App-Enhanced Brief CBT for Suicidal Inpatients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Oui Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHC-2022-0057
Record Dates: First submitted 2022-07-25; First posted 2022-08-03 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Suicidal and Self-injurious Behavior
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App-Enhanced Brief Cognitive-Behavioral Therapy (Experimental): Up to 4 in-person sessions
  Interventions: Behavioral: App-Enhanced Brief Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: App-Enhanced Brief Cognitive-Behavioral Therapy — BCBT is a cognitive-behavioral intervention designed to target core skills deficits among suicidal individuals. App-enhanced BCBT incorporates the use of a SmartPhone app during the therapy sessions.

SUMMARY:
The purpose of this study is to evaluate the feasibility of integrating Brief Cognitive-Behavioral Therapy (BCBT) counseling with a software application (app) to prevent future suicidal thoughts and behaviors.

DETAILED DESCRIPTION:
Participants will provide written informed consent. Participants will complete up to 4 sessions of BCBT (depending on length of stay) incorporating the use of a SmartPhone app. This study treatment will be completed in addition to usual care in an open trial design. Assessments will be completed at intake, discharge, and 1-, 2-, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* History of suicide attempt (lifetime) AND active ideation (with or without plan or intent) on admission
* Own and have access to their phone (iPhone or Android with capability to download apps) during their inpatient stay
* Ability to understand the nature of the study and provide written informed consent
* Willing and able to provide at least two verifiable contacts for emergency or tracking purposes
* Expected length of stay long enough to complete the entire treatment protocol

Exclusion Criteria:

* Not fluent in English
* Experiencing current mania or psychosis
* Have lifetime history of schizophrenia spectrum disorder, intellectual disability, or organic brain illness
* Inpatient treatment plan includes detox protocol or electroconvulsive therapy
* Any other psychiatric or medical condition that in the investigator's opinion would preclude informed consent or participation in the trial

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Diefenbach, PhD, Principal Investigator — Anxiety Disorders Center, Institute of Living; David Tolin, PhD, Principal Investigator — Anxiety Disorders Center, Institute of Living
Locations (1):
- Anxiety Disorders Center, Institute of Living, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Started | 4
Completed | 1
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.00 (2.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Suicidal Ideation Baseline [Mean (Standard Deviation); unit: score on a scale] — The Adult Suicidal Ideation Questionnaire (ASIQ) assesses the frequency of suicidal ideation. The ASIQ contains 25 items rated on a 0-6 scale. Items are added together for a total score ranging from 0 to 150. Higher scores indicate more frequent suicidal ideation. Means and standard deviations will be reported utilizing all available data.
  score on a scale | 82.00 (58.09)

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction at Discharge
Description: The Client Satisfaction Questionnaire (CSQ) contains 8 multiple choice items and assesses the acceptability and satisfaction of the study treatment. Items are rated from 1 to 4. Items are added together for a total score ranging from 8 to 32 with higher numbers representing greater satisfaction with the treatment. The mean and standard deviation for the CSQ total score will be reported utilizing all available data.
Time Frame: Assessed at completion of inpatient treatment (average of 16 days from admission)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Number analyzed (Participants) | 3
score on a scale | 29.00 (3.61)

2. Primary Outcome: App Usability at Discharge
Description: The System Usability Scale (SUS) contains 10 items assessing the usability of digital technology. Items are rated from 1 to 5, with higher numbers representing stronger agreement with usability statements. Scores can range from 0 to 100, with higher scores reflecting better outcomes, meaning increased usability of the technology. The mean and standard deviation for the SUS will be reported utilizing all available data.
Time Frame: Assessed at completion of inpatient treatment (average of 16 days from admission)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Number analyzed (Participants) | 3
score on a scale | 95.00 (4.33)

3. Primary Outcome: Frequency of Suicide Attempts
Description: Frequency (percentage) of participants who made a suicide attempt over the entire follow-up period
Time Frame: 3 months post-discharge from inpatient unit
Measure: Count of Participants; unit: Participants
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Number analyzed (Participants) | 3
Participants | 0

4. Primary Outcome: Suicidal Ideation Baseline
Description: The Adult Suicidal Ideation Questionnaire (ASIQ) assesses the frequency of suicidal ideation. The ASIQ contains 25 items rated on a 0-6 scale. Items are added together for a total score ranging from 0 to 150. Higher scores indicate more frequent suicidal ideation. Means and standard deviations of the total score will be reported utilizing all available data.
Time Frame: Baseline (before receiving BCBT intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Number analyzed (Participants) | 4
score on a scale | 82.00 (58.09)

5. Primary Outcome: Suicidal Ideation at Discharge
Description: as for outcome 4
Time Frame: Assessed at completion of inpatient treatment (average of 16 days from admission)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Number analyzed (Participants) | 3
score on a scale | 46.67 (19.14)

6. Primary Outcome: Suicidal Ideation 1 Month
Description: as for outcome 4
Time Frame: 1 month after discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Number analyzed (Participants) | 3
score on a scale | 21.00 (7.21)

7. Primary Outcome: Suicidal Ideation 2 Months
Description: as for outcome 4
Time Frame: 2 months after discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Number analyzed (Participants) | 1
score on a scale | 25.00 (0)

8. Primary Outcome: Suicidal Ideation 3 Months
Description: as for outcome 4
Time Frame: 3 months after discharge
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
Number analyzed (Participants) | 1
score on a scale | 45.00 (0)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the participants' inpatient admission (average length of stay 16 days) and 3 months after their discharge from the inpatient unit.
Arm/Group | App-Enhanced Brief Cognitive-Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | App-Enhanced Brief Cognitive-Behavioral Therapy (N=4)
Side effects from new medication (Psychiatric disorders) | 1 (1) — Increased anxiety and shaking associated with new medication (lithium) during inpatient stay
ED visit (Psychiatric disorders) | 1 (1) — ED visit for medication refill only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT05486091/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT05486091/ICF_001.pdf